CLINICAL TRIAL: NCT02731313
Title: Evaluation of Human HER-2 Status in Gastric and Gastro-Oesophageal Junction Cancer.
Brief Title: Human Epidermal Growth Factor Receptor 2 (HER-2) Status in Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27940
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma: Tumor samples with histologically confirmed gastric or GEJ adenocarcinoma, any stage, were collected and analyzed. No study visits or interventions were planned.
  Interventions: Biological: Trastuzumab

INTERVENTIONS:
Biological: Trastuzumab — Trastuzumab was not administered in this study. This study informs future trastuzumab treatment decisions.
  Other Names: Herceptin

SUMMARY:
The primary objective is to evaluate the concordance between human epidermal growth factor receptor 2 (HER2) status determined by the participating laboratory and by the centralized laboratory. HER2 status of samples was tested by the participating laboratories (investigator's choice of immunohistochemistry [IHC] and in situ hybridization [ISH] methods) and by the centralized laboratories (IHC using the 4B5 anti-HER antibody and Silver ISH). Positive HER2 status was defined as a score of IHC3+ or IHC2+/ISH+.

ELIGIBILITY:
Inclusion Criteria:

* Tumor samples with histologically confirmed gastric or gastro-esophageal junction (GEJ) adenocarcinoma, any stage
* Samples with sufficient tumor material for centralized analysis
* Samples fixed and embedded in paraffin (formalin-fixed paraffin-embedded tissue [FFPET] samples).

Exclusion Criteria:

- Fixatives not allowed: Bouin's solution

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor samples from participants with gastric and gastro-esophageal junction (GEJ) carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- France (16):
  - Amiens
  - Besançon
  - Boulogne-Billancourt
  - Brest
  - Clichy
  - Douai
  - La Tronche
  - Le Pontet
  - Marseille
  - Montpellier
  - Nantes
  - Paris
  - Pessac
  - Reims
  - Rennes
  - Rouen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 448 tumor specimens originating from 420 participants were assessed for inclusion in the study. Of these 448 specimens, 54 were excluded from analysis. 394 tumor specimen were included in the study which were derived from a population of 367 participants. This population (n=367) is reported in this study.
Period: Overall Study
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Started | 367
Completed | 367
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma Samples: Tumor samples with histologically confirmed gastric or GEJ adenocarcinoma, any stage, were collected and analyzed. No study visits or interventions were planned
  Trastuzumab: Trastuzumab was not administered in this study. This study informs future trastuzumab treatment decisions.
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma Samples
Number analyzed (Participants) | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 254

OUTCOME MEASURES:

1. Primary Outcome: Simple Kappa Coefficient of Human Epidermal Growth Factor Receptor 2 (HER-2) Status Between Local and Centralized Laboratory Assessments
Description: Positive HER-2 status was defined as either immunohistochemistry (IHC) score of 3+ or IHC score 2+/in situ hybridization (ISH) score +, as per the trastuzumab Summary of Product Characteristics (SPC). The HER-2 status in tumor specimens was determined using the pathologist's choice of IHC and ISH techniques in local laboratories, and using IHC 4B5 and silver ISH (SISH) in centralized laboratories. The kappa coefficient was used to evaluate the true concordance between the HER-2 status determined by local and centralized laboratories. The kappa coefficient value was interpreted according to the Landis and Koch classification as follows: a) less than (<) 0: less than chance agreement, b) 0.01-0.20: slight agreement, c) 0.21-0.40: fair agreement, d) 0.41-0.60: moderate agreement, e) 0.61-0.80: substantial agreement, and f) 0.81-0.99: almost perfect agreement.
Time Frame: At enrollment
Population: The specimens' population is defined as all specimens for which at least one IHC and/or ISH test was done in the centralized laboratory, without any reasons for exclusion.
Measure: Number (95% Confidence Interval); unit: kappa coefficient
Units Other Than Participants: Tumor specimens
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Number analyzed (Participants) | 367
Number analyzed (Tumor specimens) | 394
kappa coefficient | 0.69 [0.60 to 0.78]
Statistical Analysis 1: Comparison: Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma; Rationale for the determination of the number of samples:The following hypotheses were considered: two-sided risk alpha = 5%, power (1 - beta) = 90%, a success rate (rate of positive HER-2 status) = 17%, null hypothesis (H0): kappa coefficient = 0.90. 359 samples would allow determining a first estimate of the 0.90 coefficient of correlation kappa. The total number of samples, which had to be included in this study was 395, considering a 10% rate of non-evaluable samples; Test type: Non-Inferiority or Equivalence — Null hypothesis (H0): kappa coefficient = 0.90; p = 0.7436, Kappa-test p-value, 2 sided

2. Secondary Outcome: Cancer Characteristics: Percentage of Participants With Initial Location of Adenocarcinoma in Stomach Versus Esogastric Location
Time Frame: At enrollment
Population: The participants' sub-population being all participants from the specimen population, which is defined as all specimens for which at least one IHC and/or ISH test was done in the centralized laboratory, without any reasons for exclusion. Here, 'n' is number of participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Number analyzed (Participants) | 366
percentage of participants
  Stomach | 59.6
  Esogastric junction | 40.4

3. Secondary Outcome: Cancer Characteristics: Percentage of Participants With Samples in Each of the Histologic Type Lauren's Classifications, Including Diffuse Type, Intestinal and Mixed
Description: The Lauren classification is based on examination of histologic specimens under the microscope and divides adenocarcinoma of the stomach into 3 types: 1) Diffuse type: tumor cells are poorly differentiated, behave aggressively and tend to scatter throughout the stomach (rather than form glands). This type metastasizes to other parts of the body much quicker than intestinal type tumors, 2) Intestinal type: tumor cells are well differentiated, grow slowly and tend to form glands, 3) Mixed type: this type is made up of both intestinal and diffuse types.
Time Frame: At enrollment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Number analyzed (Participants) | 365
percentage of participants
  Diffuse type | 29.6
  Intestinal type | 54.8
  Mixed type | 9.6
  Non-evaluable | 0.3
  Other types | 5.8

4. Secondary Outcome: Cancer Characteristics: Percentage of Participants With Samples in Each of the Tumor-Node-Metastasis (TNM) Stages
Description: The TNM stage system includes information about the size of the primary tumor (T), whether the cancer has spread to nearby lymph nodes (N) and whether the cancer has metastasized to other parts of the body (M). In the T classification TX indicates that the main tumor cannot be measured, T1, T2, T3 and T4 refer to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. In the N classification NX indicates that the cancer in nearby lymph nodes cannot be measured, N0 indicates that there is no cancer in nearby lymph nodes, N1, N2 and N3 refer to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer. In the M classification MX indicates that the metastasis cannot be measured, M0 indicates that the cancer has not spread to other parts of the body and M1 indicates that the cancer has spread to other parts of the body.
Time Frame: At enrollment
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Number analyzed (Participants) | 366
percentage of participants
  T1 | 9.8
  T2 | 8.2
  T3 | 26.0
  T4 | 12.6
  Tx | 43.4
  N0 | 23.0
  N1 | 10.7
  N2 | 12.0
  N3 | 9.0
  Nx | 45.4
  M0 | 18.6
  M1 | 5.5
  Mx | 76.0

5. Secondary Outcome: Weighted Kappa Coefficient Between Immunohistochemistry (IHC) 4B5 and Silver in Situ Hybridization (SISH) Techniques for HER-2 Testing in Centralized Laboratories
Description: Positive HER-2 status was defined as either immunohistochemistry (IHC) score of 3+ or IHC score 2+/in situ hybridization (ISH) score +, as per the trastuzumab Summary of Product Characteristics (SPC). The HER-2 status in tumor specimens was determined using IHC 4B5 and silver ISH (SISH) in centralized laboratories. The weighted kappa coefficient was used to evaluate the true concordance between the HER-2 status determined by IHC 4B5 and SISH. The weighted kappa coefficient value was interpreted according to the Landis and Koch classification as follows: a) less than (<) 0: less than chance agreement, b) 0.01-0.20: slight agreement, c) 0.21-0.40: fair agreement, d) 0.41-0.60: moderate agreement, e) 0.61-0.80: substantial agreement, and f) 0.81-0.99: almost perfect agreement.
Time Frame: At enrollment
Population: The specimens' population is defined as all specimens for which at least one IHC and/or ISH test was done in the centralized laboratory, without any reasons for exclusion. Here, 'n' is number of specimens with available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: weighted kappa coefficient
Units Other Than Participants: Specimens
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Number analyzed (Participants) | 366
Number analyzed (Specimens) | 393
weighted kappa coefficient | 0.64 [0.56 to 0.72]

ADVERSE EVENTS:
Description: Adverse events were not collected for this study.
Arm/Group | Gastric and Gastro-Esophageal Junction (GEJ) Carcinoma
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.